CLINICAL TRIAL: NCT05585151
Title: High-Resolution Assessment of Extracranial Plaques in a Multiple Centers Evolocumab Randomized Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hu Bo, head of Neurology Department, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HERALD
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Atherosclerosis
Keywords: atherosclerosis; plaque burden; Evolocumab; High-Resolution assessment; OCT
MeSH Terms: conditions — Intracranial Arteriosclerosis; Atherosclerosis | interventions — evolocumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evolocumab treatment group (Experimental): Evolocumab treatment, 1ml：140mg, every 2 weeks, for 26 weeks
  Interventions: Drug: Evolocumab 140 MG/ML
- Intensive statin treatment group (Active Comparator): Atorvastatin 40mg/day or rosuvastatin 20mg/day, for 26 weeks
  Interventions: Drug: Intensive statin treatment

INTERVENTIONS:
Drug: Evolocumab 140 MG/ML — Evolocumab 140mg, subcutaneous injection, every 2 weeks, for 26 week, total 13 times
  Arms: Evolocumab treatment group
Drug: Intensive statin treatment — Intensive statin could choose either Atorvastatin 40mg/day or Rosuvastatin 20mg/day, for 26 weeks
  Arms: Intensive statin treatment group

SUMMARY:
This study intends to explore the therapeutic effect of PCSK9i Evolocumab on atherosclerotic plaques in cerebral arteries (including carotid and vertebral arteries) compared with intensive statin treatment, and monitor the pathological properties of carotid/vertebral artery plaques with OCT technology. At the same time, three-dimensional ultrasound and high-resolution magnetic resonance are used to explore the new mechanism of pathological changes of cerebral atherosclerotic plaques in a multidimensional manner.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, regardless of sex;
2. Cerebrovascular angiography examination was performed, and the imaging characteristics were consistent with: 1) The stenosis degree of internal carotid artery (starting from C1 segment) or vertebral artery (starting from vertebral artery to V4 segment) was 20%-69%; 2) The target vessel for imaging has not undergone or intends to undergo revascularization and must be available for OCT imaging catheter;
3. Participants who understand and sign the informed consent form voluntarily.

Exclusion Criteria:

1. Intolerant to both atorvastatin and rosuvastatin;
2. History of major surgery or endovascular treatment within 3 months prior to the screening period;
3. Arterial stenosis or occlusion not caused by atherosclerosis, such as arterial dissection, moya-moya disease, vasculitis, radiation vascular disease, or fibromuscular dysplasia;
4. Abnormal liver function (ALT > 3 times the upper limit of normal);
5. Renal dysfunction (glomerular filtration rate (eGFR) <45 mL/min/1.73m2 at screening);
6. Thrombocytopenia (PLT<100G/L);
7. The expected survival time is not more than 6 months;
8. Other known serious life-threatening disease (such as hematologic disease, malignancy), unstable vital signs or need for continuous monitoring, or moribund state during screening;
9. Patients have been included in other studies that conflict with this study;
10. Known sensitivity to any of the products or components to be administered during dosing;
11. Pregnant, breastfeeding or planning pregnancy, and other conditions that the investigator considers the patient unsuitable for enrollment;
12. Other conditions that the investigator considered inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes of the thickness of fibrous cap of artery plaque measured by OCT | 27 Weeks ± 7 days
  Changes of the thickness of fibrous cap of artery plaque measured by OCT

SECONDARY OUTCOMES:
Changes of the lipid arc of artery plaque measured by OCT | 27 Weeks ± 7 days
  Changes of the lipid arc of artery plaque measured by OCT
Changes of the minimum lumen area (MLA) measured by OCT | 27 Weeks ± 7 days
  Changes of the minimum lumen area (MLA) measured by OCT
Changes of lumen area stenosis measured by OCT | 27 Weeks ± 7 days
  Changes of lumen area stenosis measured by OCT
Changes of the number of microvessels measured by OCT | 27 Weeks ± 7 days
  Changes of the number of microvessels measured by OCT
Changes of the presence and extension of macrophages measured by OCT | 27 Weeks ± 7 days
  Changes of the presence and extension of macrophages measured by OCT
Changes of the calcium aggregation measured by OCT | 27 Weeks ± 7 days
  Changes of the calcium aggregation measured by OCT
Changes of arterial plaque volume measured by OCT | 27 Weeks ± 7 days
  Changes of arterial plaque volume measured by OCT
Changes of lipid necrotic core of arterial plaque measured by OCT | 27 Weeks ± 7 days
  Changes of lipid necrotic core of arterial plaque measured by OCT
Changes of LDL-C levels | 27 Weeks ± 7 days
  Changes of LDL-C levels
Changes of the thickness of minimum fibrous cap of artery plaque measured by 3D-ultrasound | 27 Weeks ± 7 days
  Changes of the thickness of minimum fibrous cap of artery plaque measured by 3D-ultrasound
Changes of arterial plaque volume measured by 3D-ultrasound | 27 Weeks ± 7 days
  Changes of arterial plaque volume measured by 3D-ultrasound
Changes of Lipid necrotic core of arterial plaque measured by 3D-ultrasound | 27 Weeks ± 7 days
  Changes of Lipid necrotic core of arterial plaque measured by 3D-ultrasound
Changes of the thickness of minimum fibrous cap of artery plaque measured by High resolution magnetic resonance | 27 Weeks ± 7 days
  Changes of the thickness of minimum fibrous cap of artery plaque measured by High resolution magnetic resonance
Changes of arterial plaque volume measured by High resolution magnetic resonance | 27 Weeks ± 7 days
  Changes of arterial plaque volume measured by High resolution magnetic resonance
Changes of Lipid necrotic core of arterial plaque measured by High resolution magnetic resonance | 27 Weeks ± 7 days
  Changes of Lipid necrotic core of arterial plaque measured by High resolution magnetic resonance
Correlation between arterial plaque and new risk factors for cardiovascular and cerebrovascular diseases (serum hsCRP, other markers, etc.) | 27 Weeks ± 7 days
  Correlation between arterial plaque and new risk factors for cardiovascular and cerebrovascular diseases (serum hsCRP, other markers, etc.)

OTHER OUTCOMES:
Occurrence of ischemic vascular events | 27 Weeks ± 7 days
  Occurrence of ischemic vascular events, such as TIA, acute cerebral infarction, acute myocardial infarction, etc.
Adverse events/serious adverse events | through study completion, an average of 6 months
  Adverse events/serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bo Hu, Doctor, Study Chair — Union Hospital, Tongji Medical College, Huahzong University of Science and Technology; Candong Hong, Doctor, Principal Investigator — Union Hospital, Tongji Medical College, Huahzong University of Science and Technology; Lei Zhang, Doctor, Principal Investigator — Union Hospital, Tongji Medical College, Huahzong University of Science and Technology; Quanwei He, Doctor, Principal Investigator — Union Hospital, Tongji Medical College, Huahzong University of Science and Technology; Jiehong Wu, Doctor, Principal Investigator — Union Hospital, Tongji Medical College, Huahzong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China